CLINICAL TRIAL: NCT04534088
Title: A Virtual-reality Based Approach to Improve Behavioral Weight Management Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VH-CP
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Behavioral Weight Loss plus Non-Weight-Related VR app (Active Comparator): The VR tool was an attention control and was not weight related.
  Interventions: Behavioral: Standard Behavioral Weight Loss plus Non-Weight-Related VR app
- Standard Behavioral Weight Loss plus Weight-Related VR app (Experimental): The Intervention's VR tool was designed to enable practice of behavioral skills taught in weekly group meetings, including managing social and home environmental cues for eating and activity.
  Interventions: Behavioral: Standard Behavioral Weight Loss plus Weight-Related VR app

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss plus Non-Weight-Related VR app — Standard Behavioral Weight Loss Program
  Arms: Standard Behavioral Weight Loss plus Non-Weight-Related VR app
Behavioral: Standard Behavioral Weight Loss plus Weight-Related VR app — Standard Behavioral Weight Loss plus Weight-Related VR app
  Arms: Standard Behavioral Weight Loss plus Weight-Related VR app

SUMMARY:
A pilot randomized trial was done to test the feasibility integrating virtual reality (VR) into standard behavioral weight loss treatment.

DETAILED DESCRIPTION:
Participants with overweight or obesity are randomly assigned to a 4-week Standard Behavioral Weight Loss plus Non-Weight-Related VR app (i.e., Control Group) or Standard Behavioral Weight Loss plus Weight-Related VR app (i.e., Intervention Group). The Intervention's VR tool was designed to enable practice of behavioral skills taught in weekly group meetings, including managing social and home environmental cues for eating and activity.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant Adults (age > 18 years) Overweight or obesity (BMI ≥ 25) Able to speak and read in English. Available on Thursday evenings Have an iPhone 6 or higher

Exclusion Criteria:

Self-reported serious psychological problems or medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Intervention Satisfaction | 4 weeks
  Participant satisfaction ratings of virtual reality scenarios on a scale where 1 = very dissatisfied to 4 = very satisfied

SECONDARY OUTCOMES:
Proportion of participants retained | 4 weeks
  Number of participants who complete the final assessment divided by the number of participants enrolled at baseline

OTHER OUTCOMES:
weight loss | 4 weeks
  weight loss from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Phelan, PhD, Principal Investigator — Cal Poly Dept. KPH
Locations (1):
- Cal Poly, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phelan S, Peruvemba S, Levinson D, Stulberg N, Lacy A, Legato M, Werner JP. Feasibility of a virtual reality-based approach to improve behavioral weight management outcomes. Pilot Feasibility Stud. 2021 Jun 22;7(1):129. doi: 10.1186/s40814-021-00865-5. PMID 34158129